CLINICAL TRIAL: NCT02963415
Title: Concurrent Aerobic Exercise and Cognitive Training to Prevent Alzheimer's in At-risk Older Adults
Brief Title: Concurrent Aerobic Exercise and Virtual Reality Cognitive Training
Acronym: VRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1610M98324
Record Dates: First submitted 2016-11-08; First posted 2016-11-15 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Preclinical Alzheimer's Disease
Keywords: Subjective memory complaint
MeSH Terms: interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Cognitive Training (Experimental): Exergame to stimulate cognition
  Interventions: Behavioral: Exergame

INTERVENTIONS:
Behavioral: Exergame — Participants will take part in the exergame, 3 times a week for a month. The session will start for 30-35 minutes of cycling on recumbent stationary cycles in session 1 and progress to moderate intensity for 50 minutes a session. Participants will do warm-up and cool-down activities before and after cycling. While cycling, participants will be playing virtual reality based games. An exercise interventionist will supervise the sessions and monitor participant's conditions and responses to ensure safety.

SUMMARY:
The study will implement and test a unique Virtual Reality Cognitive Training (VRCT) combined with concurrent cycling on a recumbent stationary cycle, also known as exergame that seamlessly integrates specific cognitive tasks into a virtual environment and is synchronized with cycling to promote cognition.

DETAILED DESCRIPTION:
The proposed project will implement and test a unique Virtual Reality Cognitive Training (VRCT) combined with concurrent cycling on a recumbent stationary cycle, also known as exergame that seamlessly integrates specific cognitive tasks into a virtual environment and is synchronized with cycling to promote cognition. Cycling through an interesting virtual environment will motivate and engage the older adult to participate in the exercise, and VRCT could augment cycling's effects on cognition. The purpose of this project is to demonstrate the feasibility and efficacy of the exergame intervention on cognition through two phases. In Phase I, a prototype of the VRCT exergame will be developed, followed by a feasibility testing using a single-group mixed methods design. In Phase II a more fully-featured version of the VRCT exergame will be developed followed by a an RCT which will randomize subjects on a 2:1:1 allocation ratio to 3 parallel groups (exergame:cycling only:attention control). Mixed methods will be used to assess outcomes in both phases.

ELIGIBILITY:
Inclusion Criteria:

1. Cognitive complaint (defined as answering yes to the question "Do you feel that your memory or thinking skills have gotten worse recently?)
2. Not engaging in aerobic exercise or cognitive training >2 days/week, 30 minutes a session in the past 3 months;
3. Age 65 years and older

Exclusion Criteria:

1. Resting heart rate > 100 or < 50 beats/min;
2. Dementia (self-report, diagnosis, or scoring <18 on the modified Telephone Interview for Cognitive Status;
3. Neurological or major psychiatric disorder since memory problem;
4. Significant diseases, symptoms, or other factors that make exercise unsafe
5. Current enrollment in another intervention study

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of the exergame development | Baseline to 3 months
  development of the exergame prototype by 3 months

SECONDARY OUTCOMES:
Cycling adherence rate | 3-6 months
  ≥70% subjects adhere to the cycling dose
VCRT adherence rate | 3-6 months
  ≥70% subjects adhere to the cognitive training dose
Usability and satisfaction with the exergame | 3-6 months
  Participants report acceptable usability and satisfaction with the exergame

CONTACTS AND LOCATIONS:
Overall Officials: Fang Yu, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No